CLINICAL TRIAL: NCT01319630
Title: The Effect of Three Different Fluids(Albumin 5%, Normal Saline, HES 130 kD) on Microcirculation in Severe Sepsis/Septic Shock Patients Using Sidestream Dark Field (SDF) Microscopy and Near-Infrared Spectroscopy (NIRS) Analysis
Brief Title: The Effect of Three Different Fluids(Albumin 5%, Normal Saline, Hydroxyethyl Starch 130 kD) on Microcirculation in Severe Sepsis/Septic Shock Patients
Status: Completed | Type: Observational
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Farid Sadaka, MD, Principal Investigator, Mercy Research
Other Study IDs: 11-007
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Severe Sepsis; Septic Shock; Microcirculation
Keywords: sepsis; microcirculation; saline; crystalloid; colloid; albumin; hydroxyethyl starch
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Saline: patients with severe sepsis/septic shock randomized to receive 1500 cc of Normal saline bolus as the resuscitation fluid.
  Interventions: Device: Sidestream Dark Field (SDF); Device: Near Infrared Spectroscopy (NIRS)
- Albumin: patients with severe sepsis/septic shock randomized to receive 500 cc of Albumin 5% bolus as the resuscitation fluid.
  Interventions: Device: Sidestream Dark Field (SDF); Device: Near Infrared Spectroscopy (NIRS)
- HES: patients with severe sepsis/septic shock randomized to receive 500 cc of Hydroxyethyl starch (HES 130kD) bolus as the resuscitation fluid.
  Interventions: Device: Sidestream Dark Field (SDF); Device: Near Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Sidestream Dark Field (SDF) — SDF will be applied to the sublingual microvascular network with a 5X objective providing a 167X magnification.
  After the removal of saliva and other secretions using gauze, the device will be gently applied (without any pressure) on the lateral side of the tongue, in an area approximately 1.5-4 cm from the tip of the tongue. Five sequences of 20 secs each from different adjacent areas will be recorded using a computer and a video card and stored under a random number for later analysis. This will be done at baseline and then 1 hour after Fluid bolus.
  Other Names: SDF ((Microscan; Microvision Medical, Amsterdam, the Netherlands)
Device: Near Infrared Spectroscopy (NIRS) — Tissue oxygen saturation (StO2) will be measured by a tissue spectrometer, a noninvasive tool, which uses reflectance mode probes to measure scattering light reflected at some distance from where the light is transmitted into the tissue. The NIRS probe will be placed on the skin of the thenar eminence and a sphygmomanometer cuff will be wrapped around the arm over the brachial artery. After a 3-min period to stabilize the NIRS signal, arterial inflow will be stopped (VOT) by inflating the cuff to 50 mmHg above the systolic arterial pressure. After 3 min of ischemia, cuff pressure will be released, and StO2 recorded continuously for another 3 min period (reperfusion period=Reactive Hyperemia).This will be done at baseline and then 1 hour after fluid bolus.
  Other Names: NIRS (InSpectra Model 650, Hutchinson Technology, Hutchinson, Minn.)

SUMMARY:
Major microvascular blood flow alterations have been documented in patients with severe sepsis. It was also demonstrated that the microcirculation improved in survivors of septic shock but failed to do so in patients dying from acute circulatory failure or with multiple organ failure after shock resolution. Early, effective fluid resuscitation is a key component in the management of patients with severe sepsis and septic shock with the goal of improving tissue perfusion. The best fluid in this early resuscitation phase has been and still is under debate. The aim of this study is to evaluate the effect of Three different Fluids(Albumin 5%, Normal Saline, HES 130 kD) on microcirculation in severe sepsis/septic shock patients using Sidestream Dark Field (SDF) Microscopy and Near-Infrared Spectroscopy (NIRS) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients will be enrolled within 24 hrs of onset of severe sepsis/septic shock with an indication for fluid bolus administration.

Exclusion Criteria:

* Liver cirrhosis
* shock from other causes
* Oral injuries (precluding SDF imaging)
* Severe peripheral vascular disease, dialysis fistula, or mastectomies precluding safe forearm occlusion
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to the Intensive Care Unit with diagnosis of sepsis.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Microcirculatory perfusion and flow variables | 1 hour after fluid bolus
  obtained by Sidestream Dark Field (SDF) microscopy
Muscle tissue oxygenation and oxygen consumption | 1 hour after fluid bolus
  using Near Infrared spectroscopy (NIRS)
change in microcirculatory and oxygenation variables | 1 hour after fluid bolus compared to baseline microcirculatory and oxygenation variables
  obtained by both SDF and NIRS

CONTACTS AND LOCATIONS:
Overall Officials: Farid G Sadaka, MD, Principal Investigator — Mercy Hospital St. Louis
Locations (1):
- St. John's Mercy Medical Center, St Louis, Missouri, United States